CLINICAL TRIAL: NCT06450379
Title: The Impact of Pneumococcal and Malaria Vaccines on Bacterial Resistance, Febrile Illness and Antibiotic Usage in Young Children in Malawi
Brief Title: Impact of Vaccines on Antimicrobial Microbial Resistance
Acronym: IVAR
Status: Completed | Type: Observational
Sponsor: Malawi Liverpool Wellcome Programme (Other)
Collaborators: Wellcome Trust (Other); University of Liverpool (Other); Kamuzu University of Health Sciences (Other); Liverpool School of Tropical Medicine (Other); University of Oxford (Other); Wellcome Sanger Institute (Other)
Responsible Party: Principal Investigator, Thoko Kapalamula, Local Principal Investigator, Malawi Liverpool Wellcome Programme
Other Study IDs: P.01/21/3249
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 13-valent pneumococcal conjugate vaccine (PCV13): 3+0 group: Children less than 3 years having received 1 dose of (PCV13) at 6, 10 and 14 weeks of age
- 13-valent pneumococcal conjugate vaccine (PCV13): 2+1 booster group: Children less than 3 years having received 1 dose of (PCV13) at 6 and 14 weeks of age and a booster at 9 months of age
- RTS,S/AS01 Vaccine-exposed: Children less than 3 years having received RTS,S/AS01 vaccine
- RTS,S/AS01 Vaccine-non exposed: Children less than 3 years having not received RTS,S/AS01 vaccine

SUMMARY:
Vaccination is a potentially critical component of efforts to arrest development and dissemination of antimicrobial resistance (AMR), though little is known about vaccination impact within low-income and middle-income countries. This study will evaluate the impact of vaccination on reducing carriage prevalence of resistant Streptococcus pneumoniae and extended spectrum beta-lactamase-producing Escherichia coli and Klebsiella species. We will leverage two large ongoing cluster-randomised vaccine evaluations in Malawi assessing; first, adding a booster dose to the 13-valent pneumococcal conjugate vaccine (PCV13) schedule, and second, introduction of the RTS,S/AS01 malaria vaccine.

Six cross-sectional surveys will be implemented within primary healthcare centres (n=3000 users of outpatient facilities per survey) and their local communities (n=700 healthy children per survey): three surveys in Blantyre district (PCV13 component) and three surveys in Mangochi district (RTS,S/AS01 component). We will evaluate antibiotic prescription practices and AMR carriage in children ≤3 years. For the PCV13 component, surveys will be conducted 9, 18 and 33 months following a 3+0 to 2+1 schedule change. For the RTS,S/AS01 component, surveys will be conducted 32, 44 and 56 months post-RTS,S/AS01 introduction. Six health centres in each study component will be randomly selected for study inclusion. Between intervention arms, the primary outcome will be the difference in penicillin non-susceptibility prevalence among S. pneumoniae nasopharyngeal carriage isolates in healthy children. The study is powered to detect an absolute change of 13 percentage points (ie, 35% vs 22% penicillin non-susceptibility).

This study has been approved by the Kamuzu University of Health Sciences (Ref: P01-21-3249), University College London (Ref: 18331/002) and University of Liverpool (Ref: 9908) Research Ethics Committees. Parental/caregiver verbal or written informed consent will be obtained prior to inclusion or recruitment in the health centre-based and community-based activities, respectively. Results will be disseminated via the Malawi Ministry of Health, WHO, peer-reviewed publications and conference presentations.

DETAILED DESCRIPTION:
Type of research study: A series of community and health centre based cross-sectional surveys

Problem: Pneumonia is a leading cause of child mortality globally and Streptococcus pneumoniae a leading cause of lower respiratory tract infections (LRTI) in under-fives. Malaria remains endemic in much of sub- Saharan Africa, commonly causing febrile illness in children and despite substantial progress with control programmes, Malaria continues to be a leading cause of child mortality. Vaccination is therefore an attractive solution.

Vaccines are thought to be crucial to Anti-Microbial Resistance (AMR) control but their impact on AMR may be more complex than originally thought. Both the direct and indirect impacts of vaccine on AMR require a systematic evaluation. In collaboration with the Malawi Ministry of Health, we are commencing two funded, regulatory approved, cluster-randomised evaluations of vaccines that target two of the commonest causes of febrile illness and life-threatening disease in children under 5 years in Africa: pneumococcal invasive infection, and malaria. This study will leverage two large funded cluster- randomised vaccine evaluations (13-valent Pneumococcal Conjugate Vaccine (PCV13) schedule change of 3+0 to 2+1 and RTS,S/AS01 (trade name Mosquirix) malaria vaccine introduction). We will assess the selective effects of pneumococcal and malaria vaccines on antibiotic resistance, febrile illness and antibiotic usage in children <3 years.

Hypothesis: Extending vaccine-mediated protection against Streptococcus pneumoniae through a 3+0 to 2+1 schedule change will be associated with a reduction in the prevalence of S. pneumoniae carriage isolates with increased AMR in children <3 years. The introduction of the malaria vaccine will reduce the frequency of healthcare attendances resulting in antibiotic prescription, reduce the prevalence of Extended spectrum beta-lactamases (ESBL) Escheriquia coli or Klebsiellae in the stool of children <3 years, and change the upper respiratory tract resistome profile in children <3years.

Aim: To establish the direct and indirect selective effects of pneumococcal and malaria vaccines on antibiotic resistance, febrile illness, and antibiotic usage in young children in Malawi.

Objectives:

1. To establish the antibiotic resistance profile of S. pneumoniae carriage isolates from children <3 years following a PCV13 schedule change that extends protection (2+1 vs. 3+0), or the introduction of malaria vaccine (RTS,S/AS01)
2. To assess the frequency of febrile illness and antibiotic use in children <3 years after PCV13 schedule change or malaria vaccine introduction
3. To investigate change in the upper respiratory tract resistome in children <3 years after PCV13 schedule change or malaria vaccine introduction.

Methodology: Three cross sectional sampling surveys shall be conducted (1) shortly following introduction of PCV13 2+1, followed by surveys 18 and 33 months after introduction, and (2) for RTS,S/AS01 2.5 years, 3 years and 3.5 years after introduction, in clusters defined through two large cluster-randomised vaccine evaluation studies. These will include the collection of nasopharyngeal and rectal swabs, and the completion of an Individual questionnaire on febrile illness episodes, malaria Rapid Diagnostic Test (RDT) use, and medicine usage with a focus on antibiotics. Additionally, we will monitor antimicrobial prescription and febrile illness at health centre level within the communities where the study will take place by conducting Health Centre (HC) Audits. These will consist of very brief anonymized "exit interviews" to randomly selected Outer-Patient Department (OPD) users, in which we will record information on the relevant vaccine (either RTS,S/AS01 or PCV13), malaria RDT (as a proxy for febrile illness) and medicine prescription

Expected Results Nasopharyngeal and rectal swabs obtained from participants will be tested for the presence of S. pneumoniae, and E. coli and Klebsiella isolates respectively. Bacterial isolates will be tested for the presence of AMR genes, and resistance profiles will be analysed in relation to their association to either the introduction of the RTS,S/AS01 vaccine or the PCV13 schedule change, and in the context of antibiotic prescription and usage for febrile illness episodes.

Outcome Measures:

Primary: The antibiotic resistance profile of S. pneumoniae carriage isolates from children <3 years following a PCV13 schedule that extends protection (2+1 vs. 3+0) or the introduction of malaria vaccine (RTS,S/AS01)

Secondary:

1. The frequency of febrile illness and antibiotic use in children <3 years after PCV13 schedule changeor malaria vaccine introduction.
2. The stool carriage of ESBL E. coli or Klebsiella in children <3 years after PCV13 schedule change or malaria vaccine introduction.
3. The change in the upper respiratory tract resistome in children <3 years after PCV13 schedule change or malaria vaccine introduction.

Population Eligibility: For the PCV13 schedule change, each cross-sectional survey shall recruit children between the ages of 4-9 months for the baseline survey, and 15 and 24 months old for the subsequent surveys, resident in Blantyre district, recruited from the community. For RTS,S/AS01, each cross-sectional survey shall recruit children between the ages of 18 and 36 months, resident in Mangochi, recruited from the community. Anonymous audits of RDT and medicine use in children <3 years attending a subset of HCs for investigation of ill health will also be conducted.

Findings' dissemination: Investigators will seek timely publication in peer-reviewed journals. Partial results and interim analyses will be shared with the Malawi Ministry of Health (MoH), and other relevant policymakers and decision-making stakeholders. Partial and final findings will be presented at the College of Medicine (COM Research Dissemination Day, Malawi-Liverpool Wellcome Trust (MWL) research in progress meetings and international scientific conferences. A copy of all published materials and reports will be shared with College of Medicine Research Ethics Committee (COMREC), and the Malawi College of Medicine Library.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residence in Blantyre (PCV cohort) or Mangochi (RTS,S/AS01 cohort)
* Parent/legal guardian consent
* Evidence of having received an initial 2 or 3 doses of the PCV13 vaccine (survey 1) or the full PCV13 schedule (surveys 2 and 3: Either 2+1 or 3+0 depending on cluster) or full initial (+/- booster) course of the RTS,S/SA01 vaccine (in Mangochi intervention cluster).

Exclusion Criteria:

* Current tuberculosis (TB) treatment
* Terminal illness (Defined as a condition that cannot be cured and it is likely to lead to the individual's death)
* Having received antibiotic treatment <14 days before study enrolment
* Hospitalisation for pneumonia <14 days before study enrolment
* Presence of gross respiratory tract pathology

For the HC audits, we will request to review the health information from attendees that comply with the following characteristics:

* <3 years of age
* HC attendance for investigation and/or treatment of ill health

Ages: 5 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under the age of 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 13200 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The antibiotic resistance profile of S. pneumoniae carriage isolates from children <3 years following a PCV13 schedule that extends protection (2+1 vs. 3+0) or the introduction of malaria vaccine (RTS,S/AS01) | less than 3 years
  This outcome measure focused on assessing the antibiotic resistance profile of Streptococcus pneumoniae isolates obtained from nasal or throat swabs of children under the age of 3. We compared two different vaccination schedules for the pneumococcal conjugate vaccine (PCV13) through a 3+0 dosing schedule and through a 2+1 dosing schedule (two primary doses followed by a booster). Additionally, the impact of the introduction of the malaria vaccine (RTS,S/AS01) on the antibiotic resistance profile of S. pneumoniae isolates was evaluated. This outcome measure aimed to determine whether different vaccination schedules or the introduction of the malaria vaccine influenced the prevalence or patterns of antibiotic resistance in S. pneumoniae, a common bacterial pathogen associated with respiratory infections in young children.

SECONDARY OUTCOMES:
The frequency of febrile illness and antibiotic use in children <3 years after PCV13 schedule change or malaria vaccine introduction. | less than 3 years
  aimed to understand how these interventions affect child health. This involved gathering data on illness and antibiotic use against changes in schedules to analyze any changes. The findings will inform public health strategies for improving child health outcomes.
The stool carriage of ESBL E. coli or Klebsiella in children <3 years after PCV13 schedule change or malaria vaccine introduction. | less than 3 years
  This is significant for understanding the impact of these interventions on bacterial resistance patterns. Here, we examed stool samples from children on different vaccine schedule change or malaria vaccine introduction to determine if there were any changes in the prevalence of ESBL E. coli or Klebsiella. Analyzing this data provided insights into how these interventions affect bacterial colonization in young children.
The change in the upper respiratory tract resistome in children <3 years after PCV13 schedule change or malaria vaccine introduction. | less than 3 years
  Examined how the upper respiratory tract's collection of antibiotic resistance genes, known as the resistome, changes in children under 3 years old following a shift in the PCV13 vaccine schedule or malaria vaccine introduction.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Heyderman, Professor, Study Chair — University College, London
Locations (1):
- Malawi Liverpool Wellcome Programme, Blantyre, Malawi